CLINICAL TRIAL: NCT02687997
Title: Prevalence of Sleep Apnea in a Lung Cancer Screening Cohort Meeting NLST Criteria
Brief Title: Prevalence of Sleep Disordered Breathing in a Lung Cancer Screening Cohort
Acronym: SAILS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, LUIS SEIJO MACEIRAS, Attending Physician, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: InsitutoFJD
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Sleep Apnea Hypopnea Syndrome; COPD; Emphysema; Lung Cancer
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnostic (Experimental): Patients enrolled in lung cancer screening subjected to a sleep study.
  Interventions: Other: poligraphy
- Contro (No Intervention): Patients enrolled in lung cancer screening not included in the diagnostic intervention arm

INTERVENTIONS:
Other: poligraphy — Sleep study
  Arms: Diagnostic

SUMMARY:
Prospective study of sleep disordered breathing in a lung cancer screening cohort.

DETAILED DESCRIPTION:
The proposed study is a prospective single arm study evaluating the prevalence of sleep disordered breathing in a cohort of lung cancer screening patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-75.
* > 30 pack years tobacco exposure.
* Enrolled in lung cancer screening program.

Exclusion Criteria:

* Inability or unwillingness to undergo a home sleep study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep apnea | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain